CLINICAL TRIAL: NCT03155841
Title: Reducing HIV Vulnerability Through A Multilevel Life Skills Intervention For Adolescent Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Michigan (Other); Emory University (Other); University of North Carolina (Other); George Washington University (Other); San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U01MD011274 (NIH)
Record Dates: First submitted 2017-05-10; First posted 2017-05-16 (Actual); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: HIV Infections; Sexually Transmitted Diseases; Sexual Behavior; Adolescent Behavior; Homosexuality
Keywords: Prevention; Internet; Adolescence; LGBT; Sexuality
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Sexual Behavior; Adolescent Behavior; Homosexuality; Sexuality | interventions — Community Resources

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Life Skills Coaching (Experimental): Participants in the experimental arm will receive access to HIV prevention and life skills content, including opportunities for goal setting, a directory of local resources in their community, and the ability to discuss their goals with Youth Navigators through a video-chat function.
  Interventions: Behavioral: Life Skills Coaching
- Community Resources (Active Comparator): Participants in the control arm will receive access to a directory of local resources in their community.
  Interventions: Behavioral: Community Resources

INTERVENTIONS:
Behavioral: Life Skills Coaching — The investigators designed the intervention to help participants increase their HIV risk awareness, promote self-appraisal and increase motivation for engaging in prevention services, problem solving barriers to accessing care, and locating culturally-sensitive providers. Intervention content is customized based on participants' socio-demographic characteristics and geographic location.
  Arms: Life Skills Coaching
Behavioral: Community Resources — The investigators will provide a resource locator as the attention-control condition. The resource locator provides a list of health (e.g., HIV testing) and social (e.g., support groups) resources across study regions.
  Arms: Community Resources

SUMMARY:
The investigators propose to deliver and test a life skills intervention targeting the key domains that fuel HIV disparities among adolescent (ages 13-18) same-sex attracted men in the United States. This RCT will yield important information regarding the delivery of a developmentally-appropriate HIV prevention program that reaches racial/ethnic and socioeconomically diverse sample of adolescent men across four regions in the United States.

DETAILED DESCRIPTION:
From 2000-2010, the annual number of new HIV diagnoses among MSM aged 13-24 years old more than doubled. There are stark racial and ethnic disparities in the incidence of new HIV infections among YMSM; 13- 24 year old racial and ethnic minority MSM now represent a rapidly growing share of all new HIV infections. Although the likelihood of HIV acquisition is greater at older ages, many of the cognitive and behavioral risk factors that contribute to the risk of HIV infection rates develop in adolescence. As adolescent MSM (AMSM; 13-18 years old) begin to develop and express gender and sexual identities, to experiment and begin sexual behaviors, and to begin to establish a sense of self, there is the opportunity to parallel this period of growth with targeted, tailored interventions that equip AMSM with the life skills they need to reduce their vulnerability to HIV risk and to establish the life skills necessary to manage risk. The investigators developed a mobile-friendly WebApp intervention focused on life skills training with links to local resources. In the proposed activities, the investigators will adapt the life skills intervention for four U.S regions heavily impacted by HIV, and revise the content to include materials that are age-appropriate for 13 to 18 year-olds. Given the role that stigma and social isolation plays in the lives of many AMSM, the investigators also propose to embed a peer-to-peer motivational interviewing component, allowing participants to access motivational interviewing counseling via VSee video-chat. With a large and diverse sample (n=500), the investigators will test the efficacy of the intervention, now referred to as iCON+, on cognitive and behavioral HIV-related outcomes using a two-arm randomized control design. In addition, the investigators examine whether structural characteristics in a region (e.g., race/ethnicity segregation, HIV prevalence) influence the efficacy of the proposed intervention.

The following Specific Aims are proposed:

1. Adapt a multilevel, online life skills intervention to address HIV vulnerability among AMSM living in four heavily impacted regions constituting diverse racial/ethnic and geographic areas (Chicago-Detroit; Atlanta-Washington, DC; Memphis- New Orleans; San Francisco-San Diego) in the US.
2. Test the efficacy of our intervention, as compared to a delayed intervention condition, to improve cognitive (e.g., comfort discussing sexuality; HIV prevention attitudes, norms, self-efficacy, behavioral intentions) and behavioral (e.g., condom use, HIV testing, PrEP use) factors using a prospective RCT design.
3. Examine the differential efficacy of our intervention in improving psychosocial mediators (e.g., personal competency) associated with our outcomes; and,
4. Examine how socio-ecological determinants at the individual (e.g., race/ethnicity, urbanity) and regional (e.g., socioeconomic disadvantage, HIV prevalence) level are associated with intervention efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Assigned a male sex at birth and identifying as male at time of enrollment,
2. Be between the ages of 13-18 (inclusive),
3. Speak and read English,
4. Report same-sex attractions and/or behaviors,
5. Live in one of the zip codes of the 109 counties included in this trial,
6. Access to internet

Exclusion Criteria:

1. Being assigned a sex other than male at birth,
2. Identifying as a gender other than male at time of enrollment,
3. Being younger than 13 or older than 18 years of age,
4. Not speaking and reading English,
5. Reporting no same-sex attractions and/or behaviors,
6. Living outside of the 109 counties included in the four regions selected for this trial,
7. Currently incarcerated,
8. No access to internet.

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Life Skills Coaching | Community Resources
Started | 300 | 300
Completed | 297 | 296
Not Completed | 3 | 4
Not completed — Protocol Violation | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Life Skills Coaching | Community Resources | Total
Number analyzed (Participants) | 300 | 300 | 600
Age, Customized [Count of Participants; unit: Participants]
  Ages 13-14 | 41 | 37 | 78
  Ages 15-16 | 136 | 128 | 264
  Ages 17-18 | 123 | 135 | 258
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 300 | 300 | 600
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 120 | 104 | 224
  Not Hispanic or Latino | 180 | 196 | 376
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 11 | 20
  Asian | 28 | 36 | 64
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 62 | 62 | 124
  White | 121 | 109 | 230
  More than one race | 54 | 45 | 99
  Unknown or Not Reported | 26 | 35 | 61
Same-sex sexual behaviors [Count of Participants; unit: Participants] — Participants reporting prior lifetime sexual behavior with a male partner
  Participants | 139 | 136 | 275

OUTCOME MEASURES:

1. Primary Outcome: Confidence to Engage in HIV Prevention Behaviors When Engaging in Receptive Anal Sex Over Time
Description: The investigators will measure HIV prevention self-efficacy over time, using a 4-point scale (1=Very Easily; 2=Easily; 3=Somewhat Easily; 4=Not Easily) where lower scores indicate a better outcome.
Time Frame: 6-month, 12-month
Population: Number analyzed in follow-up periods differ from the enrolled sample due to missing data resulting from attrition in follow-up periods. Only those participants who were measured at a given follow-up period contributed to the data reported in the table.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Life Skills Coaching | Community Resources
Number analyzed (Participants) | 240 | 257
units on a scale
  6 Month Follow-up | 1.72 (.69) | 1.71 (.69)
  12 Month Follow-up: number analyzed (Participants) | 230 | 247
  12 Month Follow-up | 1.73 (.72) | 1.72 (.71)

2. Primary Outcome: HIV Knowledge Over Time
Description: The investigators will measure HIV prevention knowledge over time using 13 True or False statements (0=Incorrect; 1=Correct) regarding HIV transmission. Scores can range from 0 to 13, where higher scores indicate a better outcome.
Time Frame: 6-month, 12-month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Life Skills Coaching | Community Resources
Number analyzed (Participants) | 238 | 260
score on a scale
  6 Month Follow-up | 7.86 (3.23) | 7.99 (2.84)
  12 Month Follow-up: number analyzed (Participants) | 227 | 249
  12 Month Follow-up | 8.33 (3.00) | 8.23 (2.98)

3. Secondary Outcome: Number of Participants Engaging in 1+ Same-Sex Sexual Partnerships
Description: The investigators will estimate participants' likelihood of engaging in one or more same-sex sexual partnerships during follow-up periods.
Time Frame: 6-month, 12-month
Measure: Count of Participants; unit: Participants
Arm/Group | Life Skills Coaching | Community Resources
Number analyzed (Participants) | 300 | 300
Participants
  6 Month Follow-Up | 78 | 84
  12 Month Follow-Up | 81 | 88

4. Secondary Outcome: Number of Participants Engaging in HIV Testing Behavior
Description: The investigators will estimate the number of participants who tested for HIV two or more times over the trial period.
Time Frame: 12-month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Life Skills Coaching | Community Resources
Number analyzed (Participants) | 189 | 199
Participants | 19 | 30

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 12 months
Arm/Group | Life Skills Coaching | Community Resources
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300 | 0/300
Other Adverse Events (participants affected / at risk) | 2/300 | 3/300
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Life Skills Coaching (N=300) | Community Resources (N=300)
HIV Infection (Infections and infestations) | 2 (2) | 3 (3) — Count of participants who self-disclosed a change in their HIV status after testing for HIV during the study period

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03155841/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT03155841/SAP_001.pdf
  • Informed Consent Form (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT03155841/ICF_002.pdf